CLINICAL TRIAL: NCT02823184
Title: Endoplasmic Reticulum Stress and Resistance to Treatments in Ph-negative Myeloproliferative Neoplasms
Acronym: PhiNESS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2014/27
Record Dates: First submitted 2016-06-24; First posted 2016-07-06 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia
Keywords: Myeloproliferative neoplasms; Endoplasmic reticulum stress
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: ET or PV patients diagnosed before acceleration phase and treated by hydroxyurea with a follow up period of at least 6 months following treatment start, with a RNA sample of total leukocytes before start of treatment available
  Interventions: Biological: RNA sample of total leukocytes before start of treatment

INTERVENTIONS:
Biological: RNA sample of total leukocytes before start of treatment — RNA sample of total leukocytes before start of treatment

SUMMARY:
The aim of this study is to evaluate the endoplasmic reticulum stress markers as predictive for response to hydroxyurea in polycythemia vera (PV) and essential thrombocythemia (ET).

DETAILED DESCRIPTION:
The recent discovery of calreticulin mutations in myeloproliferative neoplasms point to the unexpected role of the endoplasmic reticulum biology in the pathophysiology in these diseases. Otherwise, the association of endoplasmic reticulum stress with solid cancers, in particular in resistance to chemotherapy, is well documented, contrary to hematological malignancies. The study aims to evaluate endoplasmic reticulum stress markers as predictors for the response to hydroxyurea in polycythemia vera and essential thrombocythemia patients. The main objective is to correlate endoplasmic reticulum stress (defined as splicing of XBP1 above 30%) to the rate of complete response after 6 months according to the 2009 ELN criteria. This is an observational retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* ET or PV patients diagnosed before acceleration phase and treated by hydroxyurea with a follow up period of at least 6 months following treatment start.
* Diagnosis criteria of PV :

  * WHO criteria of PV with :

    * Acquired JAK2V617F mutation > 5%
    * Absence of evident cause of secondary polycythemia
* Diagnosis criteria of ET :

  * Platelet count > 450 G/L
  * Absence of PV or Chronic Myeloid Leukemia
  * Bone marrow biopsy preferred but not necessary in absence of reactional causes (CRP and ferritin levels normal) and/or presence of acquired JAK2V617F, CALR exon 9 or MPL exon 10
* Availability of RNA sample of total leukocytes before start of treatment.

Exclusion Criteria:

In absence of clonality marker, presence of secondary cause of :

* Thrombocytosis :

  * Inflammatory syndrom (CRP or SV increased)
  * Iron deficiency (decreased ferritin level or increased soluble transferrin receptor level)
* Polycythemia :

  * Increased or normal level of EPO in context of :

    * Hypoxia, respiratory insufficiency
    * Sleep apnea syndrome
    * Hyperaffin hemoglobin
* Absence of treatment by hydroxyurea
* Treatment by anagrelide, P32, pipobroman, interferon without subsequent hydroxyurea treatment.
* Concommitant treatment by other cancer chemotherapy (in a context of solid cancer for example).
* Diagnostic during transformation to acute leukemia
* Treatment by hydroxyurea during less than 6 months
* Bad observance of the cytotoxic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Polycythemia Vera or Essential Thrombocythemia
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2019-04-27 (Actual); Study Completion 2019-04-27 (Actual)

PRIMARY OUTCOMES:
To correlate endoplasmic reticulum stress (defined as splicing of XBP1 above 30%) to the rate of complete response after 6 months according to the 2009 ELN criteria | After 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MANSIER, Doctor, Principal Investigator — University Hospital, Bordeaux
Locations (7):
- France (7):
  - Chu Angers, Angers
  - Ch de La Cöte Basque, Bayonne
  - Chu de Bordeaux, Bordeaux
  - Crlcc Bergonie, Bordeaux
  - Chu de Brest, Brest
  - Ch de Dax, Dax
  - Ch de Libourne, Libourne

IPD SHARING:
Plan to Share IPD: No